CLINICAL TRIAL: NCT03967301
Title: Prevention and Decolonization of Carbapenemase-producing Enterobacteriaceae With Probiotics
Brief Title: Prevention and Decolonization of Multidrug-resistant Bacteria With Probiotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 3738
Record Dates: First submitted 2019-02-03; First posted 2019-05-30 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Probiotics; Enterobacteriaceae Infections
Keywords: Carbapenemase-producing Enterobacteriaceae; probiotics
MeSH Terms: conditions — Enterobacteriaceae Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic isolated intestinal bacteria (active) (Experimental): Patients randomized to active arm, will consume 5ml every 12 hours per day of a suspension of probiotics (Bioflora ® Lactobacillus casei, Lactobacillus plantarum, Streptococcus faecalis y Bifidobacterium brevis) for 14 days.The content of each bottle is reconstituted up to 50 ml (10 doses) with drinking water The prescription of the intervention will be carried out and monitored through the electronic medical record. In the hospital setting, the probiotic is reconstituted by the nursing staff. If the patient is discharged before this period the patient and family will be instructed to perform the reconstitution at home.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Patients randomized to the placebo arm, will consume 5ml every 12 hours per day of a suspension of placebo for 14 days. The prescription of the intervention will be carried out and monitored through the electronic medical record.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Intervention: defined as probiotic consumption
  Arms: Probiotic isolated intestinal bacteria (active)
Dietary Supplement: Placebo — Placebo consumption. The placebo will be provided by the company that produces the probiotic.
  Arms: Placebo

SUMMARY:
This study explores the effect of probiotic administration to decrease colonization by Carbapenem resistant Enterobacteriaceae (CRE) in at-risk populations. Colonized patients will be randomized to receive probiotics or placebo for 14 days and reevaluated for colonization in follow up.

DETAILED DESCRIPTION:
The use of antibiotics is known to have significant effects on the intestinal microbiota. Studies have linked this alteration with the risk of colonization and / or infection by Carbapenem resistant Enterobacteriaceae (CRE) and / or Clostridium difficile (Cd). The impact of these microorganisms has been demonstrated, with mortality rates in inpatients of around 30-50% for patients infected with CRE and 10% in Cd. It is necessary to implement mechanisms to contain dissemination and decrease colonization, in order to prevent infections caused by such agents.

Probiotics are foods consisting of live microorganisms and could restore the balance of the microbiota and avoid colonization by multi-resistant germs. Systematic reviews have shown a protective effect of probiotics for Cd. Studies on the effect on CRE are scarce and have been related mostly to prevention of colonization. Among the probiotics obtained by bacterial fermentation technology and already available in pharmacopoeia we have Bioflora ®. The objective of this trial is to explore the effect of probiotic consumption to decrease the duration of the colonization by CRE by comparing the percentage of patients colonized with CRE after the administration of probiotics and in the untreated group.

Methodology: Randomized clinical trial, single center. Known CRE colonized patients will be randomized to consume probiotics for 14 days or placebo. Then the colonization will be evaluated by means of anal swabs as indicated by the hospital standards with a follow up of 12 weeks from the initial intervention.

If the patient is discharged, home follow-up will be scheduled to supervise the intake of the dietary supplement and the control swabs.

The expected impact is to accelerate the process of decolonization of multi-resistant germs through the administration of probiotics leading to a shorter contact isolation time in and reducing the risk of complications in CRE colonized patients.

ELIGIBILITY:
Inclusion Criteria:

* CRE- colonized patients
* adult patients in hospital (over 18 years old)
* Part of the HIBA health care plan
* CRE positive rectal swab or stool in the last 14 days

Exclusion criteria:

* Enteral route enabled (oral, nasogastric tube, gastrostomy or jejunostomy)
* Refusal to participate in the study
* Not available for weekly checks, minimum up to 12 weeks from enrollment
* Clostridium difficile active infection concomitant with CRE swab in a 14-day period days
* Neutropenia G3 or greater (less than 1000 neutrophils at the time of enrollment).
* Severe immunosuppressed at the time of recruitment according to the CDC definition (patients transplanted, HIV with CD4 <200, congenital immunodeficiencies, leukemias, lymphomas, cancer disseminated, current chemotherapy or radiotherapy, treatment with corticoids high dose:prednisone 20 mg / d> 2 weeks or immunosuppressive drugs).
* Patient with valvular prostheses
* Imminent death
* Fistula or dehiscence of the gastrointestinal tract
* Acute pancreatitis
* Patient of critical units in ileus and / or with high requirement of vasopressors (noradrenaline equal to or greater than 0.5 gammas) at the time of recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
presence of CRE in anal swab or stool culture in follow-up control: | 12 weeks
  CRE anal swab positive upon discharge, therapeutic adjustment or in-hospital death.
  ● Date of swab, therapeutic adjustment or in-hospital death.
  and within a month :
  ● Control CRE swab per month for KPC: Categorical binomial: Positive / Negative. Will be performed 30 days after enrollment and weekly for 8 weeks if positive. It will be considered negative when the patient as three consecutive negative swabs separated by a week. It will be persistently positive when during this period of follow-up at least one of the swabs is positive, total follow-up 12 weeks

SECONDARY OUTCOMES:
positive for clostridium difficile diarrhea | 12 weeks
  If a patient develops diarrhea at some point during hospitalization, screening for Cd will be performed at the attending phisician´s discretion
  If the patient has diarrhea with a positive Cd toxin and is receiving probiotic he/she should leave the study and the data for CRE will be evaluated with the last available swab at the time of the exit event (positive for clostridium difficile diarrhea).